# Clinical Performance of Two Reusable Silicone Hydrogel Contact Lenses

STUDY ID CLL949-C024

STATISTICAL ANALYSIS PLAN

NCT05766787



# Statistical Analysis Plan for CLL949-C024 Title: Clinical Performance of Two Reusable Silicone Hydrogel Contact Lenses



#### **Executive Summary:**

#### Key Objectives:

The primary objective of this study is to demonstrate noninferiority (NI) in the visual acuity (VA) at distance when wearing Alcon serafilcon A contact lenses compared to ACUVUE® OASYS with HYDRACLEAR® PLUS Technology (AOHP) contact lenses when worn in a daily wear modality.

Decision Criteria for Study Success:

Success of this study will be based on demonstration of NI in distance VA with Alcon serafilcon A contact lenses when compared to AOHP contact lenses at Week 1, using a margin of 0.05 on the logMAR scale.

# **Table of Contents**

| Sta | itistical A | nalysis Plan for CLL949-C024 | 1 |
|---|---|---|---|
| Tal | ole of Cor | ntents | 3 |
| Lis | st of Table | es | |
| Lis | st of Figur | res | |
| 1 | | OBJECTIVES AND DESIGN | |
| | 1.1 | Study Objectives | |
| | 1.2 | Study Description | |
| | 1.3 | Randomization | |
| | 1.4 | Masking | |
| | 1.5 | Interim Analysis | |
| 2 | ANALY | SIS SETS | |
| | 2.1 | Safety Analysis Sets | |
| | 2.2 | Full Analysis Set | |
| | 2.3 | Per Protocol Analysis Set | |
| 3 | SUBJEC | CT CHARACTERISTICS AND STUDY CONDUCT SUMMARIES | |
| 4 | EFFECT | ΓIVENESS ANALYSIS STRATEGY | <u></u> 9 |
| | 4.1 | Effectiveness Endpoints | 9 |
| | 4.2 | Effectiveness Hypotheses | |
| | 4.3 | Statistical Methods for Effectiveness Analyses | 13 |
| | | 4.3.1 Primary Effectiveness Analyses | |
| | 4.4 | Multiplicity Strategy | 14 |
| | 4.4 | Subgroup Analyses and Effect of Baseline Factors | |
| | 4.6 | Interim Analysis for Effectiveness | |
| 5 | | Y ANALYSIS STRATEGY | |
| 5 | 5.1 | | |
| | 5.2 | Safety Endpoints | |
| | 5.3 | Statistical Methods for Safety Analyses | |
| | 3.3 | 5.3.1 Adverse Events | |
| | | 5.3.2 Biomicroscopy Findings | |
| | | 5.3.3 Device Deficiencies | |


| 7 SAMPL | E SIZE AND POWER CALCULATIONS | 18 |
|---|---|---|
| 8 REFERI | REFERENCES | |
| 9 REVISI | ON HISTORY | 21 |
| 10 APPEN | DIX | 22 |
| m.11. 4.4 | List of Tables | |
| Table 1-1 | Study Description Summary | 5 |
| Table 10-1 | Schedule of Study Procedures and Assessments | 22 |
| | List of Figures | |
| Figure 1–1 | Study Design | 6 |

#### 1 STUDY OBJECTIVES AND DESIGN

# 1.1 Study Objectives

#### PRIMARY OBJECTIVE

The primary objective of this study is to demonstrate NI in the VA at distance when wearing Alcon serafilcon A contact lenses compared to AOHP contact lenses when worn in a daily wear modality.



# 1.2 Study Description

Key components of the study are summarized in Table 1-1.

Table 1-1Study Description Summary

| Study Design | Prospective, randomized, double masked, bilateral, crossover |
|---|---|
| Study Population | Volunteer subjects aged 18 or over who are habitual spherical |
| | soft contact lens wearers (excluding current/previous AOHP |
| | habitual lens wearers and daily disposable lens wearers), have at |
| | least 3 months of contact lens wearing experience, and who |
| | wear their habitual lenses at least 5 days per week and at least 8 |
| | hours per day. |
| | T 160 |
| | Target to complete: 168 |
| | Planned to enroll: ~ 185 |
| Number of Sites | ~ 14 |
| | US |
| Test Product | Alcon serafilcon A contact lenses (serafilcon A; LID 022821) |
| Comparator Product | ACUVUE® OASYS with HYDRACLEAR® PLUS Technology |
| | contact lenses (AOHP; senofilcon A) |
| Planned Duration of | ~ 28 days total duration (test and comparator): |
| Exposure | Test product: 14 (-0/+2) days |
| | Comparator Product: 14 (-0/+2) days |
| Visits | Visit 1: Screening/Baseline |



A study design schematic is depicted in Figure 1–1.

Week 2 follow up lens 2/Exit

Figure 1-1 **Study Design** Visit 1 Lens fitting Pre-fitting Screen / Baseline with lens fitting Informed consent Lens type 1 fitted VA, fit, surface History and CL experience 2-4 days (at least 48 hour) washout Refraction and VA Lens type 2 fitted Biomicroscopy Keratometry VA, fit, surface Visit 2 Randomization Dispense pair 1 In-office questionnaire At least 16 hrs lens wear Visit 3 Week 1 follow up lens 1 At least 16 hrs lens wear Follow-up examination Lenses on-eye Visit 4 Refraction and VA Week 2 follow up lens 1 2-4 days (at least 48 hour) washout Lenses out-of-eye Refraction and VA Visit 5 Biomicroscopy Keratometry Dispense pair 2 Lens collection At least 16 hrs lens wear Visit 6 Week 1 follow up lens 2 At least 16 hrs lens wear Visit 7

#### 1.3 Randomization

A member of the Randomization Programming group at Alcon who is not part of the study team will generate the randomized allocation schedule(s) for study lens sequence assignment. Randomization will be implemented in the Electronic Data Capture (EDC)/randomization integration system.

Qualifying subjects will be randomized in a 1:1 manner to receive treatment (lens) in crossover sequence: test product then comparator product or comparator product then test product, respectively.

| Sequence | EDC/randomization integration system | Lens Name |
|------------|--------------------------------------|-------------------------|
| Sequence 1 | LID022821/AOHP | Alcon serafilcon A/AOHP |
| Sequence 2 | AOHP/LID022821 | AOHP/Alcon serafilcon A |

#### 1.4 Masking

This study is double-masked.

#### 1.5 Interim Analysis

There are no plans to conduct an interim analysis and no criteria by which the study would be terminated early based upon statistical determination.

#### 2 ANALYSIS SETS

# 2.1 Safety Analysis Sets

Safety analyses will be conducted using the safety analysis set on a treatment-emergent basis. As such, the safety analysis set will include all subjects/eyes exposed to any study lenses evaluated in this study.

For treatment-

emergent safety analyses, subjects/eyes will be categorized under the actual study lenses exposed in the corresponding lens sequence.

Adverse events occurring from the time of informed consent but prior to first exposure to study lenses will be summarized in subject listings.

#### 2.2 Full Analysis Set



#### 2.3 Per Protocol Analysis Set

The per protocol (PP) analysis set is a subset of FAS and excludes all data/subjects that have met any of the critical deviation or evaluability criteria identified in the Deviations and Evaluability Plan (DEP).

# 3 SUBJECT CHARACTERISTICS AND STUDY CONDUCT SUMMARIES

The following tables will be presented:

- Subject Disposition by Lens Sequence
- Analysis Sets by Lens
- Analysis Sets by Lens Sequence
- Subject Accounting by Lens Sequence
- Demographics by Lens Sequence
- Baseline Characteristics by Lens Sequence [lens brand; lens power; lens care;
   keratometry readings; Best Corrected
   Visual Acuity (BCVA); habitual lens wear and rewetting drops usage]

Subject accounting and demographics tables will be summarized on the safety, full and per protocol analysis datasets. Baseline characteristics will be summarized on the full and per protocol analysis datasets.

In addition, the following subject listings will be provided:

- Listing of Subjects Excluded from Protocol Defined Analysis Sets
- Listing of Lens Sequence Assignment by Investigator

• Listing of Subjects Discontinued from Study

#### 4 EFFECTIVENESS ANALYSIS STRATEGY



All effectiveness analyses will be carried based on the randomization assignment.

Continuous variables will be summarized using the number of observations, mean, standard deviation (SD), median, minimum, and maximum, as well as confidence intervals (CIs) or confidence limits where applicable. Categorical variables will be summarized with frequencies and percentages from each category.

All data obtained in evaluable subjects/eyes will be included in the analysis. No imputation for missing values will be carried out for the primary and key exploratory effectiveness analyses.

For all planned inferential analyses, alternative models/methods may be considered if convergence cannot be achieved. Furthermore, if significant carryover effects are noted (confounded with sequence effect), results will be examined by period to ensure the overall conclusion is valid.

A listing of select effectiveness data will also be provided.

# 4.1 Effectiveness Endpoints

#### **Primary Effectiveness Endpoint**

The primary endpoint is distance VA with study lenses at Week 1, collected for each eye in logMAR.

• Time to questionnaire completion (hours or minutes, as applicable)

# 4.2 Effectiveness Hypotheses

#### **Primary Effectiveness**

The null and alternative hypotheses are formulated in terms of the predefined margin of 0.05 for noninferiority:

$$\begin{aligned} &H_0: \ \mu_{(T)} - \mu_{(C)} \geq 0.05 \\ &H_a: \ \mu_{(T)} - \mu_{(C)} \leq 0.05 \end{aligned}$$

where  $\mu_{(T)}$  and  $\mu_{(C)}$  denote the mean distance VA at Week 1 for Alcon serafilcon A and AOHP, respectively, on the logMAR scale.





#### 4.3 Statistical Methods for Effectiveness Analyses

#### **4.3.1** Primary Effectiveness Analyses

A mixed effects repeated measures model will be utilized to test these hypotheses. The model will include terms for lens, period, sequence, visit (Dispense, Week 1, Week 2), and lens by visit interaction. Within subject correlation due to eye and crossover will also be accounted for in the model. Lens difference (Alcon serafilcon A minus AOHP) and the corresponding one-sided 95% upper confidence limit (UCL) will be computed at Week 1. Noninferiority will be declared if the UCL is less than 0.05.

Document ID: Status: Approved, Version: 1.0 V-CLN-0038497 Approved Date: 03 Mar 2023


#### 4.4 Multiplicity Strategy

The primary effectiveness endpoint of distance VA will be tested at one-sided  $\alpha = 0.05$  for NI and will serve as the gatekeeper for subsequent testing of the key effectiveness endpoints.

#### 4.5 Subgroup Analyses and Effect of Baseline Factors

It is not expected that demographics or baseline characteristics will have an impact on study results in this study. No subgroup analyses are planned.

#### 4.6 Interim Analysis for Effectiveness

No interim analysis is planned for the effectiveness endpoints.

#### 5 SAFETY ANALYSIS STRATEGY

The focus of the safety analysis will be a comprehensive descriptive assessment of occurrence of adverse events as well as the other listed parameters. Therefore, no inferential testing will be done for the safety analysis.

# 5.1 Safety Endpoints

The safety endpoints are:

- AEs
- Biomicroscopy findings
  - Limbal hyperemia
  - o Bulbar hyperemia
  - Corneal staining
  - Conjunctival staining
  - Palpebral conjunctival observations
  - o Corneal epithelial edema
  - o Corneal stromal edema
  - Corneal vascularization
  - Conjunctival compression/indention
  - o Chemosis
  - Corneal infiltrates
  - Other findings

Device Deficiencies

# 5.2 Safety Hypotheses

There are no formal safety hypotheses in this study. The focus of the safety analysis will be a comprehensive descriptive assessment of safety endpoints listed in Section 5.1.

#### 5.3 Statistical Methods for Safety Analyses

The analysis set for all safety analyses is defined in Section 2.1. Baseline will be defined as the last measurement prior to exposure to study lenses. For biomicroscopy data, baseline will be defined as Visit 2 for Period 1 and Visit 5 for Period 2. Safety variables will be summarized descriptively.

#### **5.3.1** Adverse Events

The applicable definition of an AE is in the study protocol. All AEs occurring from when a subject signs the informed consent to the time of their study exit will be accounted for in the reporting.

Presentation of AEs will be separated into pre-treatment AEs, between-treatment AEs, and treatment-emergent AEs as defined below:

- Pre-treatment: an event that occurs after signing informed consent but prior to exposure to study lenses
- Between-treatment: an event that occurs one day after last exposure to Period 1 study lenses but prior to exposure of Period 2 study lenses.
- Treatment-emergent: an event that occurs from first exposure to Period 1 study lenses until subject exits from the study, excluding those classified as between-treatment

The following tables and supportive listings will be provided:

- Incidence of All Ocular Treatment-Emergent Adverse Events
- Incidence of Ocular Serious Treatment-Emergent Adverse Events
- Incidence of Ocular Significant Nonserious Treatment-Emergent Adverse Events
- Incidence of All Nonocular Treatment-Emergent Adverse Events
- Incidence of Nonocular Serious Treatment-Emergent Adverse Events
- Listing of All Ocular Treatment-Emergent Adverse Events
- Listing of All Nonocular Treatment-Emergent Adverse Events

- Listing of All Ocular Pre-Treatment Adverse Events
- Listing of All Nonocular Pre-Treatment Adverse Events
- Listing of All Ocular Between-Treatment Adverse Events
- Listing of All Nonocular Between-Treatment Adverse Events

#### 5.3.2 Biomicroscopy Findings

The following tables and supportive listings will be provided:

- Frequency and Percentage for Biomicroscopy Findings by Visit
- Incidence of Increased Severity by 2 or More Grades in Biomicroscopy Findings

Status: Approved, Version: 1.0

Approved Date: 03 Mar 2023

- Listing of Subjects With Other Biomicroscopy Findings
- Listing of Subjects With Conjunctival Compression/Indentation or Chemosis
- Listing of Subjects With Increased Severity by 2 or More Grades in Biomicroscopy Findings
- Listing of Subjects with Infiltrates

#### **5.3.3** Device Deficiencies

The following tables and supportive listings will be provided:

- Frequency of Treatment-Emergent Device Deficiencies
- Listing of Treatment-Emergent Device Deficiencies
- Listing of Device Deficiencies Prior To Treatment Exposure

#### 7 SAMPLE SIZE AND POWER CALCULATIONS

Sample size calculation is based on a prior clinical study ( which evaluated performance of Alcon serafilcon A and AOHP.



Status: Approved, Version: 1.0 Approved Date: 03 Mar 2023  Document ID: V-CLN-0038497

# 8 REFERENCES

Not applicable.

# 9 REVISION HISTORY

This is the original (Version 1.0) Statistical Analysis Plan for this study. This version of the Statistical Analysis Plan is based on Version 2.0 of the study protocol.

#### 10 APPENDIX

Table 10-1 Schedule of Study Procedures and Assessments

| | | | Ler<br>(Peri | | | | Lens 2<br>(Period 2) | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Procedure/<br>Assessment | Pres<br>cree<br>ning | Visit 1<br>Screening /<br>Baseline | Visit 2 Dispense Lens 1 [2 (at least 48 hours) – 4 days after Visit 1 (Washout period with habitual spectacles only after Visit 1)] | Visit 3 Week 1 Follow-up Lens 1 [7 -0/+ 1 days after Visit 2] | Visit 4 Week 2 Follow- up Lens 1 [7 -0/+ 1 days after Visit 3)] | Visit 5 Dispense Lens 2 [2 (at least 48 hours) – 4 days after Visit 4 (Washout period with habitual spectacles only after Visit 4)] | Visit 6 Week 1 Follow-up Lens 2 [7 -0/+ 1 days after Visit 5] | Visit 7 Week 2 Follow-up Lens 2 /Exit [7 -0/+ 1 days after Visit 6)] | Early<br>Exit | Unsche<br>duled<br>Visit |
| Informed Consent | | X | 1 | | | | | | | |
| Demographics | | X | | | | | | | | |
| Medical History | | X | X | X | X | X | X | X | X | X |
| Concomitant<br>Medications | | X | X | X | X | X | X | X | X | X |
| Inclusion/ Exclusion | | X | | | | | | | | |
| Habitual lens<br>(brand, lens<br>power, lens<br>care) | | X | | | | | | | | |
| In office subjective questionnaire • Habitual lens wear and rewetting drop usage | | Х | | | | | | | | |

| | | Lens 1<br>(Period 1) | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Procedure/<br>Assessment | Pres<br>cree<br>ning | Visit 1<br>Screening /<br>Baseline | Visit 2 Dispense Lens 1 [2 (at least 48 hours) – 4 days after Visit 1 (Washout period with habitual spectacles only after Visit 1)] | Visit 3<br>Week 1<br>Follow-up<br>Lens 1<br>[7 -0/+ 1<br>days after<br>Visit 2] | Visit 4<br>Week 2<br>Follow- up<br>Lens 1<br>[7 -0/+ 1<br>days after<br>Visit 3)] | Visit 5 Dispense Lens 2 [2 (at least 48 hours) – 4 days after Visit 4 (Washout period with habitual spectacles only after Visit 4)] | Visit 6<br>Week 1<br>Follow-up<br>Lens 2<br>[7 -0/+ 1<br>days after<br>Visit 5] | Visit 7<br>Week 2<br>Follow-up<br>Lens 2<br>/Exit<br>[7 -0/+ 1<br>days after<br>Visit 6)] | Early<br>Exit | Unsche<br>duled<br>Visit |
| Keratometry | | X | (X) | (X) | (X) | (X) | (X) | (X) | (X) | (X) |
| VA w/ habitual<br>correction <sup>+</sup><br>(OD, OS,<br>logMAR<br>distance)* | | X | (A) | (A) | (A) | (A) | (A) | X | X | (X)<br>(X) |
| Manifest refraction* | | X | (X) | (X) | (X) | (X) | (X) | (X) | (X) | (X) |
| BCVA (OD, OS,<br>logMAR distance with<br>manifest refraction) | | X | (X) | (X) | (X) | (X) | (X) | (X) | (X) | (X) |
| Biomicroscopy | | X | X | X | X | X | X | X | X | X |

| | | Lens 1<br>(Period 1) | | | | Lens 2<br>(Period 2) | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Procedure/<br>Assessment | Pres<br>cree<br>ning | Visit 1<br>Screening /<br>Baseline | Visit 2 Dispense Lens 1 [2 (at least 48 hours) – 4 days after Visit 1 (Washout period with habitual spectacles only after Visit 1)] | Visit 3 Week 1 Follow-up Lens 1 [7 -0/+ 1 days after Visit 2] | Visit 4 Week 2 Follow- up Lens 1 [7 -0/+ 1 days after Visit 3)] | Visit 5 Dispense Lens 2 [2 (at least 48 hours) – 4 days after Visit 4 (Washout period with habitual spectacles only after Visit 4)] | Visit 6<br>Week 1<br>Follow-up<br>Lens 2<br>[7 -0/+ 1<br>days after<br>Visit 5] | Visit 7 Week 2 Follow-up Lens 2 /Exit [7 -0/+ 1 days after Visit 6)] | Early<br>Exit | Unsche<br>duled<br>Visit |
| Fitting of investigational products (trial assessments): (Test and Comparator)* - VA (logMAR distance) - Lens movement (Overall fit- primary and peripheral gazes) - Lens position (Centration) | | X | | | | | | | | |
| Randomization | | X | | | | | | | | |
| Dispense study lenses VA w/study lenses, (OD, OS, logMAR distance) | | | X | X | X | X | X<br>X | X | (X) | (X)<br>(X) |

| | | | Len<br>(Peri | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Procedure/<br>Assessment | Pres<br>cree<br>ning | Visit 1<br>Screening /<br>Baseline | Visit 2 Dispense Lens 1 [2 (at least 48 hours) – 4 days after Visit 1 (Washout period with habitual spectacles only after | Visit 3<br>Week 1<br>Follow-up<br>Lens 1<br>[7 -0/+ 1<br>days after<br>Visit 2] | Visit 4 Week 2 Follow- up Lens 1 [7 -0/+ 1 days after Visit 3)] | Visit 5 Dispense Lens 2 [2 (at least 48 hours) – 4 days after Visit 4 (Washout period with habitual spectacles only after | Visit 6 Week 1 Follow-up Lens 2 [7 -0/+ 1 days after Visit 5] | Visit 7 Week 2 Follow-up Lens 2 /Exit [7 -0/+ 1 days after Visit 6)] | Early<br>Exit | Unsche<br>duled<br>Visit |

| | | | Lens 1<br>(Period 1) | | | | Lens 2<br>(Period 2) | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Procedure/ | Pres | Visit 1 | Visit 2 | Visit 3 | Visit 4 | Visit 5 | Visit 6 | Visit 7 | Early | Unsche |
| Assessment | cree | Screening / | Dispense | Week 1 | Week 2 | Dispense | Week 1 | Week 2 | Exit | duled |
| | ning | Baseline | Lens 1 | Follow-up | Follow- up | Lens 2 | Follow-up | Follow-up | | Visit |
| | | | [2 (at least | Lens 1 | Lens 1 | [2 (at least | Lens 2 | Lens 2 | | |
| | | | 48 hours) – | [7 -0/+ 1 | [7 -0/+ 1 | 48 hours) – | [7 -0/+ 1 | /Exit | | |
| | | | 4 days after | days after | days after | 4 days after | days after | [7 -0/+ 1 | | |
| | | | Visit 1 | Visit 2] | Visit 3)] | Visit 4 | Visit 5] | days after | | |
| | | | (Washout | | | (Washout | | Visit 6)] | | |
| | | | period with | | | period with | | | | |
| | | | habitual | | | habitual | | | | |
| | | | spectacles | | | spectacles | | | | |
| | | | only after | | | only after | | | | |

| AEs α | X | X | X | X | X | X | X | X | X | |
|---------------------|-----|-----|-----|-----|-----|-----|---|---|-----|---|
| Device deficiencies | X | X | X | X | X | X | X | X | X | l |
| Exit Form | (X) | (X) | (X) | (X) | (X) | (X) | X | X | (X) | I |

- (X) Assessment performed as necessary, e.g., decrease of VA by 2 lines or more with investigational product (IP)
- \* Source only (source transferred to the sponsor upon request)
- α Comprehensive details of all AEs will be documented in the source records, however limited collection will be utilized in the eCRF (see MOP for details).

# Signature Page for V-CLN-0038497 v1.0



Signature Page for V-CLN-0038497 v1.0